CLINICAL TRIAL: NCT04415398
Title: Fully Integrated Drone-system for Delivery of an Automated External Defibrillator (AED) in Out-of-hospital Cardiac Arrest (OHCA) Before the Arrival of Emergency Medical Services (EMS)
Brief Title: AED-delivery Using Drones in Out-of-hospital Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: SOS Alarm Sverige AB (Unknown); Everdrone AB (Unknown)
Responsible Party: Principal Investigator, Andreas Claesson, Associate professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC1
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Drone; UAV
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Intervention Model Description: Totally n=3 AED-drones are deployed as a complement to standard care (EMS) in all cases of suspected OHCA occurring within service areas
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Delivery of automated external defibrillators using drones (Experimental): Three drone systems are setup to be deployed in suspected OHCA cases as a complement to EMS. This is a single-arm intervention evaluating feasibility in:
  * Operational feasibility (Legislation, Weather conditions, conflict in airspace)
  * Participant feasibility (Failure to respond; Dispatcher, Drone-pilot, Air traffic controller)
  * Technological feasibility (Drone technology, software, winch-system , 4G network, radio communication
  Interventions: Device: Automated flying Drone carrying an Automated external defibrillator (AED)

INTERVENTIONS:
Device: Automated flying Drone carrying an Automated external defibrillator (AED) — Totally n=3 drones are equipped with automated external defibrillators (AEDs). These drones are deployed by the dispatch centre to cases of suspected out-of-hospital cardiac (OHCA) as a complement to standard care (ambulance/EMS) over 4 months during daytime Monday to Sunday 08:00-22:00. The bystander onsite receives instructions from the dispatcher to retrieve the AED outside the house when it has been delivered by the drone. The bystander attaches the AED to the patients chest to facilitate early defibrillation.

SUMMARY:
Time to defibrillation is the most important predictor of survival in cardiac arrest. Traditional emergency medical system response is often to slow. The aim of this study is to investigate the feasibility of drone systems that delivers Automated External Defibrillators (AED) to the scene of suspected Out-of-Hospital Cardiac Arrests (OHCA).

This study will test the feasibility of real-life flights with drones carrying automated external defibrillators (AEDs) to out-of-hospital cardiac arrest (OHCA) as a complement to standard care i.e EMS

DETAILED DESCRIPTION:
We will test the feasibility of dispatching an out of sight AED-drone system to real-life OHCA in parallel with standard EMS dispatch. The study period is 5 months between May to September 2020. The study area will be covered by three individual drone systems covering some 80,000 inhabitants within the controlled airspace of Säve airport in Göteborg Sweden. Each drone system will have a flight range of six km.

The first month of the study period will be used as run-in period and the drone systems are dispatched for beyond visual line of sight (BVLOS) flights in a simulated fashion and optimized to decrease delays and to log pre-specified system variables, adherence to protocol, time delays, technological functionality, weather conditions, conflict in the airspace.

During the following 4 months June-September 2020, drones will dispatched to real-life suspected OHCA during daytime 08:00-22:00.

An EMS communication radio-unit is placed at the drone control center. In case of a suspected OHCA in the service area and will be alerted by the dispatch centre (SOS alarm) when a suspected OHCA is recognized during the 112-call.

* The dispatcher identifies a cardiac arrest in the service areas
* A pilot (from Everdrone) immediately initiates deployment protocol for the drone.
* Parallel communication is made with the air traffic control (ATC) centre in order to grant permit to deploy the drone with regards to the current weather and aviation situation.
* The drone then flies to the coordinates of the OHCA and delivers an AED at the scene using a winch system
* The AED may be attached to the patient by the bystander on scene

Development of the technology is made by Everdrone AB Göteborg and SOS Alarm AB (national dispatch organisation) and parallel applications for certificates for the individual aircraft and permits for beyond visual line of sight flights (BVLOS-flights) was granted by the Swedish Transportation board on 27 April 2020.

The drone system is operated only during daytime 08:00-22:00 when the Airport Air traffic control is open. Likewise deployment of the drone will not be made if there is a conflict in the airspace with manned aircrafts. Rainy weather or winds exceeding 8 m/s prohibits flights as well.

Feasibility is evaluated and measured from the following aspects:

1. Operational factors Weather: a) rain, b) wind c) other. Conflict in airspace: a) manned aircraft b) unmanned aircraft. Obstacles prohibiting flight or delivery: a) constructed b) natural Time from dispatch to to take- off (min:sec). Time from dispatch to arrival (min:sec). Proportions are measured out of cases with a) Take-off b) no take-off c) aborted missions (%)
2. Human resources Adherence to protocol by: a) Dispatcher b) Drone pilot c) Air traffic leader. Proportions are measured out of cases with neglected protocol prohibiting mission completion, a) no alerts b) no take off c) aborted missions (%)
3. Technological functionality Drone, winch, Network, AED, Hangar, navigational software, global positioning system precision, Dispatch centre system (CoordCOM -Dispatch centre automated alert).

Proportions are measured out of cases where technological functionality prohibited mission completion a) no take-off b) aborted missions. (%)

Adverse advents (AE) and serious adverse events (SAE) in relation to AED-drone mission /use will be logged continuously. An adverse event may be caused by drone crash or risc of injury or death due to conflict in airspace or technological impairment.

An AE is considered serious if it:

* Results in death
* Is immediately life-threatening
* Requires hospitalisation or prolongation of existing hospitalization
* Results in persistent or significant disability or incapacity

Events that are related to the patient in cardiac arrest and would be expected in patients undergoing attempted resuscitation should NOT be reported. These include:

* Death
* Hospitalisation
* Persistent or significant disability or incapacity
* Organ failure

All events categorised as serious must be reported to the study administration within 24 hours of becoming aware of the event.

ELIGIBILITY:
Inclusion Criteria:

* All suspected OHCA
* Within n=3 service areas
* Hours of operation: 08:00-22:00

Exclusion Criteria:

* Children <8 years
* Trauma
* EMS-witnessed cases

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of suspected OHCA cases (%) where the AED-drone was dispatched and accurately completed mission. | Up to 4 months
  All cases of OHCA within the three service areas where the dispatch centre alerts the drone-operator and the drone takes-off. Accurate completion of mission equals deliver an AED onsite on the ground within 50 meters from OHCA location. AEDs shall be accessible to the bystander through T-CPR instructions given by the dispatcher.

SECONDARY OUTCOMES:
Proportion of suspected OHCA with AED-drone arrival prior to ambulance | Up to 4 months
  Comparisons on proportion of units arriving first to the scene for ambulance vs AED-drone, percentages.
Time difference of drone arrival as compared to ambulance | Up to 4 months
  Time delay from dispatch to arrival (delivered AED on ground), minutes, seconds.
Proportion/numbers of attached drone delivered AEDs prior the arrival of EMS (%). | Up to 4 months
  A bystander retrieves the AED as instructed in T-CPR protocol by the dispatcher and attaches it to the patient before ambulance arrival. Percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Claesson, PhD, Principal Investigator — Centre for resuscitation science, Karolinska Institutet
Locations (1):
- Göteborg AED-drone service areas, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schierbeck S, Hollenberg J, Nord A, Svensson L, Nordberg P, Ringh M, Forsberg S, Lundgren P, Axelsson C, Claesson A. Automated external defibrillators delivered by drones to patients with suspected out-of-hospital cardiac arrest. Eur Heart J. 2022 Apr 14;43(15):1478-1487. doi: 10.1093/eurheartj/ehab498. PMID 34438449